CLINICAL TRIAL: NCT04178486
Title: Eating Behavior - Choice or Reconstruction of Past Experience? Changing Eating Behaviors of Healthy Adults Through Hypnotic Suggestions
Brief Title: Changing Eating Behaviors of Healthy Adults Through Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Comsa Loana, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phd Study
Record Dates: First submitted 2019-10-27; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Weight loss; Hypnosis; Eating Behavior; Free Will
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Feeding Behavior | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Participants were randomized in one of the four groups.
Who Masked: Participant
Masking Description: The participants were not informed in which group they are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amnesia (Experimental): Hypnosis formed from hypnotic induction (an adapted version from Barber Suggestibility Scale) together with hypnotic suggestions to experience amnesia for the food pictures they had just seen.
  Interventions: Behavioral: Hypnosis with amnesia suggestions
- Cognitive Rehearsal (Experimental): Hypnosis formed from hypnotic induction (an adapted version from Barber Suggestibility Scale) together with hypnotic suggestions about a future where they will control their eating behaviors.
  Interventions: Behavioral: Hypnosis with cognitive rehearsal suggestions
- Memory Substitution (Experimental): Hypnosis formed from hypnotic induction (an adapted version from Barber Suggestibility Scale) together with hypnotic suggestions about a past where they have always controlled their eating behaviors.
  Interventions: Behavioral: Hypnosis with memory substitution suggestions
- Control (Placebo Comparator): Hypnosis formed from only hypnotic induction (an adapted version from Barber Suggestibility Scale).
  Interventions: Behavioral: Hypnosis with induction only

INTERVENTIONS:
Behavioral: Hypnosis with amnesia suggestions — Participants received hypnotic induction with hypnotic suggestions for their eating behaviors.
  Arms: Amnesia
Behavioral: Hypnosis with cognitive rehearsal suggestions — Participants received hypnotic induction with hypnotic suggestions for their eating behaviors.
  Arms: Cognitive Rehearsal
Behavioral: Hypnosis with memory substitution suggestions — Participants received hypnotic induction with hypnotic suggestions for their eating behaviors.
  Arms: Memory Substitution
Behavioral: Hypnosis with induction only — Participants received only hypnotic induction.
  Arms: Control

SUMMARY:
There is a lot of research on weight loss. In spite of the research on the subject, obesity is a growing disease all through the world. The results of recent reviews and meta-analyzes show that psychological interventions had small effect on weight loss. The investigators propose a different approach to changing eating behaviors with relevance to weight management and hypothesize that participants in the active interventions will significantly improve their eating behaviors than the ones in the control group. The results will improve the psychological interventions for weight loss.

DETAILED DESCRIPTION:
This is a randomized clinical trial consisting of four groups. According to the concept of Free Will, the decision of action is taken before being acknowledged and is made following the reconstruction of previous experiences. It can be inhibited immediately (max 100ms) after awareness. The investigators want to intervene based on this model using hypnotic suggestions to change eating behaviors. Participants were found through social media announcements. Three groups receive one session of hypnosis with induction and different suggestions and the control group receives only induction. The eating behavior is measured through computer tasks in which participants have the option to choose pictures of food. The task is performed before, during and after hypnosis and the measurements of eating behavior are taken at all three times.

ELIGIBILITY:
Inclusion Criteria:

Both gender Healthy Adults who want to change their eating behavior

Exclusion Criteria:

Severe mental illness <18 years A diagnosed eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Eating Behavior | The intervention is delivered in one session. The outcome is measured: immediately pre intervention (0-2 min), during intervention and immediately post intervention (0-2 min).
  The number of food pictures chosen by the participant in this single session intervention. The outcome is a measure assessing a change between three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Loana T Comsa, Phd Student, Principal Investigator — Babes Bolyay University
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haggard P, Cartledge P, Dafydd M, Oakley DA. Anomalous control: when 'free-will' is not conscious. Conscious Cogn. 2004 Sep;13(3):646-54. doi: 10.1016/j.concog.2004.06.001. PMID 15336254
- [Background] Jamieson GA, Kittenis MD, Tivadar RI, Evans ID. Inhibition of retrieval in hypnotic amnesia: dissociation by upper-alpha gating. Neurosci Conscious. 2017 Apr 19;2017(1):nix005. doi: 10.1093/nc/nix005. eCollection 2017. PMID 30042839
- [Background] Gravitz, Melvin A.
- [Background] Oakley DA, Halligan PW. Hypnotic suggestion and cognitive neuroscience. Trends Cogn Sci. 2009 Jun;13(6):264-70. doi: 10.1016/j.tics.2009.03.004. Epub 2009 May 8. PMID 19428287
- [Background] Obhi, Sukhvinder S., and Patrick Haggard.
- [Background] Kuhn S, Haggard P, Brass M. Intentional inhibition: how the "veto-area" exerts control. Hum Brain Mapp. 2009 Sep;30(9):2834-43. doi: 10.1002/hbm.20711. PMID 19072994
- [Background] Wolpert DM, Ghahramani Z, Jordan MI. An internal model for sensorimotor integration. Science. 1995 Sep 29;269(5232):1880-2. doi: 10.1126/science.7569931.
- [Background] Haggard P. Human volition: towards a neuroscience of will. Nat Rev Neurosci. 2008 Dec;9(12):934-46. doi: 10.1038/nrn2497. PMID 19020512
- [Background] Libet, Benjamin.
- [Background] Terhune DB, Brugger P. Doing better by getting worse: posthypnotic amnesia improves random number generation. PLoS One. 2011;6(12):e29206. doi: 10.1371/journal.pone.0029206. Epub 2011 Dec 15. PMID 22195022
- [Background] Mendelsohn A, Chalamish Y, Solomonovich A, Dudai Y. Mesmerizing memories: brain substrates of episodic memory suppression in posthypnotic amnesia. Neuron. 2008 Jan 10;57(1):159-70. doi: 10.1016/j.neuron.2007.11.022. PMID 18184572
- [Background] Oakley DA, Halligan PW. Hypnotic suggestion: opportunities for cognitive neuroscience. Nat Rev Neurosci. 2013 Aug;14(8):565-76. doi: 10.1038/nrn3538. Epub 2013 Jul 17. PMID 23860312
- [Background] Stoeckel LE, Weller RE, Cook EW 3rd, Twieg DB, Knowlton RC, Cox JE. Widespread reward-system activation in obese women in response to pictures of high-calorie foods. Neuroimage. 2008 Jun;41(2):636-47. doi: 10.1016/j.neuroimage.2008.02.031. Epub 2008 Mar 4. PMID 18413289